CLINICAL TRIAL: NCT03611712
Title: PG2 Concurrent With Chemoradiation for Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-CP028
Record Dates: First submitted 2018-07-10; First posted 2018-08-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Fatigue; Survival; Tumor, Esophageal
Keywords: Cancer-related Fatigue; Tumor response; Survival; Chemoradiation; esophageal cancer
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCRT-PG2 arm (Experimental): Astragalus Polysaccharides 500 mg
  Interventions: Drug: Astragalus Polysaccharides 500 mg
- CCRT alone arm (No Intervention)

INTERVENTIONS:
Drug: Astragalus Polysaccharides 500 mg — PG2 Lyo. Injection 500 mg will be given on 1 week before CCRT (Week 1, PG2 Lyo. Injection 500 mg, b.i.w), during CCRT (Week 2-6, PG2 Lyo. Injection 500 mg, t.i.w for 5 weeks), and after CCRT (Week 7-8, PG2 Lyo. Injection 500 mg, t.i.w for 2 weeks)
  Other Names: PG2 Lyo. Injection 500 mg
  Arms: CCRT-PG2 arm

SUMMARY:
The primary objective of this study is to evaluate the efficacy of PG2 concurrent with concurrent chemoradiation therapy (CCRT) for relieving fatigue among locally advanced esophageal cancer patients who are under preoperative chemoradiation therapy at curative setting. This study will be designed to compare the fatigue status between two study arms patients under CCRT.

The secondary objective is to assess the efficacy of PG2 to improve the quality of life of patient during CCRT. Also, the investigators try to determine the effect of PG2 on tumor response post CCRT, disease free survival (DFS) and overall survival (OS) of patients by comparing the above outcome between the two study arms.

The mechanism of immunomodulatory of PG2 and tumor response, DFS and OS for patients with esophageal cancer treated with preoperative CCRT concurrent with or without PG2 will be investigated in add-on study.

DETAILED DESCRIPTION:
It's randomized, open-label study. Locally advanced esophageal cancer patients who give consent to participate in this study and meet all other inclusion and exclusion criteria will be eligible to enroll into this study. The eligible patients will be randomized into one of two study arms: 1) the CCRT- PG2 arm; and 2) the CCRT alone arm. All eligible patients will receive the standard preoperative CCRT during study period and standard surgery 6 weeks after completion of radiation therapy.

The primary objective of this study is to evaluate the efficacy of PG2 concurrent with CCRT for relieving fatigue. Patient's fatigue status will be measured by the BFI-T.

The secondary objective is to assess the efficacy of PG2 to improve the quality of life of patient during CCRT. Patients' quality of life will be assessed by the Functional Assessment of Cancer Therapy- General (FACT-G7 v.4). Patients' appetite will be assessed by VAS appetite score. The effect of PG2 on tumor response post CCRT, DFS and OS of patients will also be evaluated.

Peripheral blood samples and tumor biopsy samples will be collected from all subjects at screening period, during CCRT and post CCRT period to perform Immune biomarker assessment in the add-on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent form;
* The age of eligible patients should be 20-75 years old;
* Performance status of ECOG 0-1 at time of screening;
* Have Esophageal and esophagogastric junction cancer (non-cervical esophagus);
* Have stage IIB-IIIB locally advanced carcinoma of esophagus;
* Pathologically confirmed primary squamous cell carcinoma of the esophagus;
* Patient must be willing and able to complete fatigue and quality of life questionnaires.

Exclusion Criteria:

* BFI > 7 at time of screening;
* Concomitant malignancy or prior invasive malignancy unless disease free for a minimum of 2 years;
* Medical contraindications to esophagectomy;
* Female patients are pregnant or breast-feeding;
* Have inadequate bone marrow, liver, and renal function
* Uncontrolled systemic disease
* Regular steroid use as determined by investigators;
* Patients take central nervous system stimulators such as Methylphenidate within 30 days before screening;
* Patients have enrolled or have not yet completed other investigational drug trials within 30 days before screening.
* BMI < 16
* Nutrition status SGA rating C.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Fatigue by the Brief Fatigue Inventory-Taiwanese Form | Through 12 weeks
  The Brief Fatigue Inventory (BFI) has been shown to have good reliability of fatigue measurement. This instrument consists of a one-page fatigue assessment tool that contains nine items, each measuring the severity of fatigue on a 0-through-10 scale. The first three items assess current level of fatigue, and worst and usual fatigue in the preceding 24 hours. Six items assess the extent to which fatigue has interfered with different aspects of life, such as work or social relations, during the preceding 24 hours. The BFI score is calculated from the mean of completed items.

SECONDARY OUTCOMES:
Quality of life by the Functional Assessment of Cancer Therapy-General (FACT-G7 v.4) | Through 12 weeks
  FACT-G7, a rapid version of the Functional Assessment of Cancer Therapy-General (FACT-G) which is one of most validated assessment tools to evaluate health related qulaity of life (HRQoL) among cancer patients. It is a 27-item instrument containing four subscales: physical well-being (PWB), functional well-being (FWB), social/family well-being (SWB), and emotional well-being (EWB) on 0-4 scale with a recall period of the past 7 days. The scores of these items must be reversed, and then summed to a total, which is the subscale score. The higher score is presented as the better quality of life.
Visual Analog Score for appetite | Through 12 weeks
  Visual Analog Score for appetite is a single-item scale will be used to measure by A 10-cm vertical line anchored with the number 0 to indicate "no appetite" and number 10 to indicate "worst possible appetite."
Tumor response be evaluated by RECIST 1.1, irRECIST and Pathological response. | Week 11 and Week 12
Disease free survival | 2 years after the take-off day of the last patient
  Disease free survival (DFS) is defined as the time from initiation to relapse or death, whichever occurred first.
Overall survival in locally advanced esophageal cancer patients with PG2 treatment under preoperative chemoradiation therapy | 2 years after the take-off day of the last patient
  Overall survival (OS) is defined as the time from initiation to death of any cause.
The change of of biomarkers (inhibitory immune factors, dendritic cells makers, tumor-associated macrophages, immune-regulatory markers and oncogenic-mediated immune markers) will be combined to report the immune profile. | Through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chien WC Huang, MD, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (4):
- Taiwan (4):
  - Mackay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Taipei Medical University -Shung Ho Hospital, Taipei